CLINICAL TRIAL: NCT00947999
Title: Neurofeedback Treatment of Pain in Persons With SCI: Phase 1
Brief Title: Neurofeedback Treatment of Pain in Persons With Spinal Cord Injury (SCI)
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Mark Jensen, Principal Investigator, University of Washington
Other Study IDs: 36292-D Phase I; 124155-A
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Cord Injury; Pain
MeSH Terms: conditions — Spinal Cord Injuries; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Control Group: Subjects in particular group will not have a diagnosis of SCI and do not experience chronic pain. Subjects in this group will be matched roughly to subjects in the SCI chronic pain group based on age, gender and race/ethnicity.
- Subjects with SCI and Chronic Pain: Individuals recruited into this particular group will have a diagnosis of a spinal cord injury and experience pain on a daily basis with an average intensity of 4 out of 10 on a 0-10 scale.
- Subjects with SCI and No Chronic Pain: Subjects in particular group will have a diagnosis of SCI and not have chronic pain. Subjects in this group will be matched roughly to subjects in the SCI chronic pain group based on age, gender and race/ethnicity.

SUMMARY:
There has been little research on how chronic pain is related to brain activity. The purpose of this study is to learn more about pain and brain activity by finding any differences in brain activity among people who have moderate to severe chronic pain and a spinal cord injury, those who have a spinal cord injury but do not experience chronic pain, and people who have neither a spinal cord injury nor chronic pain (please note: subjects do not have to have pain to participate in this study). The information we collect will help the investigators get a better understanding of chronic pain.

DETAILED DESCRIPTION:
Research staff will record the brain activity of subjects by using an electroencephalogram (EEG), a device that measures the electrical activity in the brain through electrodes put on the scalp. There is no risk of electrical shock. Research staff will put a cap on the subject's head that has electrodes that will measure your brain activity. In addition to the electrodes in the cap, two electrode clips will be put on your ears. EEG activity will be collected for 20 minutes: subjects will have their eyes open for ten minutes, and then eyes closed for ten minutes.

Before the assessment, subjects will be asked how much pain they are currently in. Once the 20-minute assessment has ended, the research staff member will again ask subjects how much pain they are currently in, and how much pain they had during the EEG assessment. Subjects with SCI-related pain on a daily basis may also be contacted in the future to see if they want to participate in the second phase of this study that will involve learning to directly change their brain activity.

ELIGIBILITY:
Inclusion Criteria:

SCI Chronic Pain Group

1. 18 years old or older.
2. At least 12 months post-SCI.
3. Otherwise healthy (i.e., no other secondary medical complications, such as pressure ulcers, that could impact pain scores).
4. Read, write and understand English.
5. Experience SCI-related pain on a daily basis.
6. Report an average pain intensity of at least 4 on a 0-10 Numerical Scale.
7. An individual must have a worst or most significant pain problem if he/she has more than one pain problem.
8. Pain problem has lasted at least six months.

SCI No Pain Group

1. 18 years old or older.
2. At least 12 months post-SCI.
3. Otherwise healthy (i.e., no other secondary medical complications, such as pressure ulcers, that could impact pain scores).
4. Read, write and understand English.

Healthy Control Group

1. 18 years old or older.
2. Otherwise healthy (i.e., no other secondary medical complications, such as pressure ulcers, that could impact pain scores).
3. Read, write and understand English.

Exclusion Criteria:

SCI Chronic Pain Group

1. History of seizure activity or has non-normative brain activity.
2. Suicidal or paranoid thoughts.
3. Presence of traumatic brain injury or significant skull defects.
4. Exhibit moderate to severe cognitive impairment (<=20) on the TICS questionnaire.

SCI No Pain Group

1. History of seizure activity or has non-normative brain activity.
2. Suicidal or paranoid thoughts.
3. Presence of traumatic brain injury or significant skull defects.
4. Experience pain more than once a week.
5. Exhibit moderate to severe cognitive impairment (<=20) on the TICS questionnaire.

Healthy Control Group

1. History of seizure activity or has non-normative brain activity.
2. Suicidal or paranoid thoughts.
3. Presence of traumatic brain injury or significant skull defects.
4. Experience pain more than once a week.
5. Exhibit moderate to severe cognitive impairment (<=20) on the TICS questionnaire.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited primarily from a previous survey study conducted by the principal investigator, as well as a data registry maintained by the principal investigator. Individuals recruited for these studies were recruited primarily from rehabilitation clinics. Interested individuals may also learn about the study from advertisements in newsletters and magazines from consumer organizations, physician referrals, recruitment descriptions on University of Washington websites, and study brochures in clinics.
  In addition, SCI subjects participating in the study will give friends and relatives who do not have a spinal cord injury or chronic pain a brochure informing them about the study.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
EEG brain wave activity. | Recorded at time of assessment.

SECONDARY OUTCOMES:
Pain intensity before, during an after EEG assessment. | Collected at time of assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Jensen MP, Sherlin LH, Gertz KJ, Braden AL, Kupper AE, Gianas A, Howe JD, Hakimian S. Brain EEG activity correlates of chronic pain in persons with spinal cord injury: clinical implications. Spinal Cord. 2013 Jan;51(1):55-8. doi: 10.1038/sc.2012.84. Epub 2012 Jul 17. PMID 22801188